CLINICAL TRIAL: NCT04702282
Title: Population Pharmacokinetics of Ropivacaine Used for Local Infiltration Anesthesia During Primary Total Unilateral and Simultaneous Bilateral Knee Arthroplasty
Brief Title: Population Pharmacokinetics of Ropivacaine
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kirill Gromov, Associate Professor, Hvidovre University Hospital
Other Study IDs: H-16027950
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- unilateral Total knee arthroplasty: Patients receiving unilateral Total knee arthroplasty
  Interventions: Diagnostic Test: ropivacain concentration measurements
- simultaneous bilateral Total knee arthroplasty: Patients receiving simultaneous bilateral Total knee arthroplasty y
  Interventions: Diagnostic Test: ropivacain concentration measurements

INTERVENTIONS:
Diagnostic Test: ropivacain concentration measurements — Free and total plasma concentrations of ropivacaine were measured within 24 hours using liquid chromatography - mass spectrometry. A population pharmacokinetic model was built using non-linear mixed effect models

SUMMARY:
The aim of this study was to investigate the pharmacokinetics of free and total ropivacaine after unilateral and bilateral TKA. A population model was successfully built and peak free ropivacaine concentration stayed below previously proposed toxic thresholds in patients undergoing unilateral as well as bilateral TKA receiving LIA with high dose ropivacaine.

DETAILED DESCRIPTION:
Thirteen unilateral TKA and fifteen bilateral TKA patients were included in the study. All patients were operated in a well-described fast-track setup without use of drains or tourniquet.21 A standard midline skin incision with a medial para-patellar capsulotomy was used. All patients were operated with cemented CR components. In bilateral TKA cases, both knees were operated in one setting with the left knee always being operated first, and the second knee being operated sequentially in the same setting immediately following closure of the first knee. Patients undergoing unilateral TKA received spinal anesthesia with 2 mL 0.5% hyperbaric bupivacaine, whereas patients scheduled for bilateral TKA received spinal anaesthesia with 3 mL 0.5% hyperbaric bupivacaine. Local infiltration anesthesia was performed as previously described with 200 mL 0.2% ropivacaine (400 mg) mixed with 1 mL 1 mg/mL epinephrine injected periarticularly in each knee. The first 50 mL were injected into the posterior capsule, 100 mL were injected into medial, anterior and lateral structures of the knee and capsule and the final 50 mL were injected in the subcutaneous tissue. All patients were mobilized on the day of surgery and thromboembolic prophylaxis started 6-8 hours postoperatively with rivaroxaban tablets (10 mg) given once daily until discharge. No extended thromboembolic prophylaxis was given to any patient. All patient received 1 g intravenous tranexamic acid preoperatively and 1 g 3 hours postoperatively.

Preoperative blood samples were taken within a week of surgery including electrolytes, hemoglobin and serum creatinine levels. Baseline blood sample was taken just before incision of the first knee, and additional blood samples were drawn at 1, 5, 30 and 60 minutes as well as 2, 4, 8 and 24 hours after incision following unilateral TKA and at 1, 5, 30 minutes after the incision of the first knee and 0, 5 and 15 minutes after incision of the second knee as well as after 1,2, 4 8 and 24 hours (total 9 and 12 timepoints within 24 hours for unilateral and bilateral TKA, respectively). Patient demographics were recorded and included age, gender, height and weight.

Ropivacaine measurement Ropivacaine concentrations were determined in plasma samples using liquid-chromatography coupled to mass spectrometry following a fully validated method

ELIGIBILITY:
Inclusion criteria:

Patients undergoing unilateral TKA (n=13) and bilateral TKA (n=15) receiving LIA according to standard protocol.

Exclusion criteria:

Patients not receiving LIA Revision TKA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirteen unilateral TKA and fifteen bilateral TKA patients were included in the study. All patients were operated in a well-described fast-track setup without use of drains or tourniquet. A standard midline skin incision with a medial para-patellar capsulotomy was used. All patients were operated with cemented CR components. In bilateral TKA cases, both knees were operated in one setting with the left knee always being operated first, and the second knee being operated sequentially in the same setting immediately following closure of the first knee.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Free and total plasma concentrations of ropivacaine | 24 hours
  Free and total plasma concentrations of ropivacaine were measured within 24 hours using liquid chromatography - mass spectrometry

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gromov K, Grassin-Delyle S, Foss NB, Pedersen LM, Nielsen CS, Lamy E, Troelsen A, Urien S, Husted H. Population pharmacokinetics of ropivacaine used for local infiltration anaesthesia during primary total unilateral and simultaneous bilateral knee arthroplasty. Br J Anaesth. 2021 Apr;126(4):872-880. doi: 10.1016/j.bja.2020.11.038. Epub 2021 Jan 15. PMID 33455802